CLINICAL TRIAL: NCT00576147
Title: A Multi-Center Study of Near-Infrared Spectroscopy (NIRS) for Hematoma Detection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: InfraScan, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Infrascanner-052306
Record Dates: First submitted 2007-12-14; First posted 2007-12-18 (Estimated); Results first posted 2013-12-20 (Estimated); Last update posted 2018-11-07 (Actual); Status verified 2018-10

CONDITIONS: TBI (Traumatic Brain Injury)
Keywords: TBI; NIRS; Hematoma
MeSH Terms: conditions — Brain Injuries, Traumatic; Hematoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CT scan (Experimental): The standard head CT done to head trauma patients
  Interventions: Device: Infrascanner

INTERVENTIONS:
Device: Infrascanner — The main Near-Infrared spectroscopy (NIRS) head measurement

SUMMARY:
The purposes of this study are:

1. To determine the sensitivity and specificity of the Near-Infrared Spectroscopy (NIRS) measurements for identifying intracranial hematomas due to trauma.
2. To determine the reproducibility of the Near-Infrared Spectroscopy (NIRS) measurements with different operators and at different centers

DETAILED DESCRIPTION:
The principle used in identifying intracranial hematomas with Near-infrared spectroscopy (NIRS) is that extravascular blood absorbs Near-infrared light more than intravascular blood since there is a greater (usually 10-fold greater) concentration of hemoglobin in the acute hematoma then in the brain tissue where blood is contained within vessels. Therefore, the absorbance of Near-infrared light is greater (and therefore the reflected light less) on the side of the brain containing a hematoma, than on the uninjured side.

The NIRS sensor is placed successively in the left and right frontal, temporal, parietal, and occipital areas of the head and the absorbance of light at selected wavelengths is recorded. The difference in optical density in the different areas is calculated.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing a CT scan within 12 hours of their head injury. The criteria for obtaining a CT scan will be based on the standard of care, but generally all patients with a moderate or severe head injury will receive a CT scan on admission to the hospital, and only patients who undergo a CT will be enrolled into the study. The non-contrast CT will be performed according to standard methods.

Exclusion Criteria:

* 12 hours or more since injury.
* Massive scalp lacerations, avulsions, and hematomas The limitation to injury within 12 hours is necessary because as hematoma blood is metabolized, the absorbance characteristics change.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 431 (Actual)
Dates: Start 2006-07; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Robertson, MD, Principal Investigator — Professor Medical Director, The Center for Neurosurgical Intensive Care, Ben Taub Hospital, Houston, Texas
Locations (4):
- United States (4):
  - Johns Hopkins University, Baltimore, Maryland
  - University of Cincinnati, Cincinnati, Ohio
  - The Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Baylor College of Medicine, Houston, Texas

REFERENCES:
- [Background] Robertson CS, Gopinath S, Chance B. Use of near infrared spectroscopy to identify traumatic intracranial hemotomas. J Biomed Opt. 1997 Jan;2(1):31-41. doi: 10.1117/12.261680. No abstract available. PMID 23014820
- [Background] Gopinath SP, Robertson CS, Grossman RG, Chance B. Near-infrared spectroscopic localization of intracranial hematomas. J Neurosurg. 1993 Jul;79(1):43-7. doi: 10.3171/jns.1993.79.1.0043. PMID 8315468
- [Result] Robertson CS, Zager EL, Narayan RK, Handly N, Sharma A, Hanley DF, Garza H, Maloney-Wilensky E, Plaum JM, Koenig CH, Johnson A, Morgan T. Clinical evaluation of a portable near-infrared device for detection of traumatic intracranial hematomas. J Neurotrauma. 2010 Sep;27(9):1597-604. doi: 10.1089/neu.2010.1340. PMID 20568959

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Near-Infrared examinations performed on all patients within 30 minutes before the CT scan of the head and within 12 hours of their head injury
Period: Overall Study
Arm/Group | CT Scan
Started | 431
Completed | 431
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | CT Scan
Number analyzed (Participants) | 431
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 46
  Between 18 and 65 years | 333
  >=65 years | 52
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.7 (26)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 108
  Male | 323
Region of Enrollment [Number; unit: participants]
  United States | 306
  India | 125

OUTCOME MEASURES:

1. Primary Outcome: 1) Sensitivity of the Near-Infrared Spectroscopy (NIRS) Measurements for Identifying Intracranial Hematomas Due to Trauma. 2) Specificity of the Near-Infrared Spectroscopy (NIRS) Measurements for Identifying Intracranial Hematomas Due to Trauma.
Description: We will report Sensitivity and Specificity of NIRS device as compared to CT scanner to detect hematomas of more than 3.5 mL in volume and less than 2.5 cm from the surface of the brain.
  Sensitivity is the ratio between true positives to all positive measurements. Specificity is the ratio between true negatives to all negative measurements.
Time Frame: 2 years
Population: 431 Total patients enrolled; 365 total patients evaluated after 66 excluded for protocol violations; 269 Number of patients with no Intracranial Hemorrhage; 96 Number of patients with confirmed intrcranial hemorrhage; 50 Number of patients with Intracranial hemorrhage within detection limits of the device.
Measure: Number; unit: Number of participants
Arm/Group | CT Scan
Number analyzed (Participants) | 365
Number of participants
  True Positive | 44 [74.9 to 95.0]
  False Positive | 25
  True Negatives | 244
  False Negatives | 6
Statistical Analysis 1: Comparison: CT Scan; Test type: Superiority or Other; Percent Sensitivity = 88, 95% CI 2-sided [75.0 to 95.0]
Statistical Analysis 2: Comparison: CT Scan; Test type: Superiority or Other; Percent Specificity = 90.7, 95% CI 2-sided [86.4 to 93.7]

ADVERSE EVENTS:
Arm/Group | CT Scan
Serious Adverse Events (participants affected / at risk) | 0/431
Other Adverse Events (participants affected / at risk) | 0/431

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No